CLINICAL TRIAL: NCT04478331
Title: Effects of Technology-based Physical Activity Interventions for Women After Bariatric Surgery: a Three-arm Randomized Control Study
Brief Title: Effects of Technology-based Physical Activity Interventions for Women After Bariatric Surgery
Acronym: OCAPAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pr Fabienne d'Arripe-Longueville (Other)
Collaborators: Centre Hospitalier Universitaire de Nice (Other); Association Azur Sport Santé, Nice, France (Unknown)
Responsible Party: Sponsor-Investigator, Pr Fabienne d'Arripe-Longueville, University Professor CEX1 - Director of the Human Motricity Expertise Sport Health Laboratory (LAMHESS, UPR 6312) and co-director of the "Fédération de Recherche Interventions en Santé" (FRIS)., Universite Cote d'Azur
Organization: Universite Cote d'Azur (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IDRCB: 2020.A00172-37; ANR-15-IDEX-01 (Other Grant/Funding Number: ANR as part of the UCAJEDI Future Investments project)
Record Dates: First submitted 2020-07-10; First posted 2020-07-20 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Bariatric Surgery Candidate
Keywords: obesity; physical activity; information and communication technology; engagement; active lifestyle; technology-based program; eHealth; videoconferencing; mobile application
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CONTROL (No Intervention): The Control group will receive the usual care. In the physical activity (PA) field, this includes two individual motivational interviews with a PA professional, and a group workshop during the first year after BS. PA recommendations will be explained to each participant, and their achievement will be encouraged and supported during these sessions. No face-to-face PA sessions will be offered as part of the usual care.
- ACTI-VISIO (Experimental): The two PA sessions per week will be delivered via videoconferencing (developed by Mooven™). The PA program consists in tailored adapted PA sessions led by a professional specialized in adapted PA. These sessions were specifically designed to be appropriate for the population and were developed in collaboration with the authors to ensure standardization of the recommended volume of PA. The PA sessions will be given live, individually at the beginning and then in groups of four women. During sessions, the professional and the participants will interact simultaneously, and the execution of the exercises will be monitored and adapted live by the professional. To ensure the safety of the PA, a rating of perceived exertion will be requested after each session on a 10-point scale. If the RPE exceed 7, the professional specialized in adapted PA will adjust the training load. In addition to the exercises, the sessions will also include advice and tips for reaching the recommended PA level.
  Interventions: Behavioral: Technology-based physical activity interventions
- ACTI-MOBIL (Experimental): The PA sessions will be delivered by an eHealth platform (developed by BePatient™) associated with an activity bracelet. The researchers enrich PA content on the platform and ensure standardization of the recommended volume of PA. The platform consists of tips for reaching the PA level, PA questionnaires, PA feedback measured by the activity bracelet, and a video demonstration of PA sessions performed by a peer. The PA sessions are automatically broadcasted twice a week for 12 weeks. To ensure the safety of the PA, the sessions were designed to be appropriate for this population and the RPE will be measured after each session on a 10-point scale. If the RPE exceeds 7 for 3 consecutive sessions, the training load will be adjusted. The platform will also include a variety of content, including dietary tips, obesity-related facts, information about surgery, and frequently asked questions.
  Interventions: Behavioral: Technology-based physical activity interventions

INTERVENTIONS:
Behavioral: Technology-based physical activity interventions — The technology groups will receive a PA program for 12 weeks. These PA programs will be given twice a week and include: 5-10 minutes of warm-up, 20-40 minutes of aerobic exercise and muscle strengthening via circuit training composed of 8-10 exercises with 8-12 repetitions per exercise for 2-3 series, and 5-10 minutes of stretching. In addition, advice and counseling will be given about walking activities to achieve the recommendations.
  Arms: ACTI-MOBIL; ACTI-VISIO

SUMMARY:
Regular physical activity (PA) is essential throughout bariatric surgery (BS) management, especially for the long-term maintenance of weight loss. To optimize physical activity counseling and monitoring, the use of technology seems appropriate and effective. A recent meta-analysis provided proof of efficacy for mobile technology to increase physical activity or weight loss in the short term. Videoconferencing may also be effective, especially as it reduces the barriers related to face-to-face physical activity interventions. Both technologies (mobile and videoconferencing) seem particularly interesting for bariatric surgery management, but their long-term effects on physical activity maintenance are unknown. Moreover, the mechanisms underlying their effectiveness, such as technology acceptability and motivational processes, have not been examined.

The purpose of this study is to determine the effects of two technology-based (mobile technology and videoconferencing) PA programs after BS compared to standard care and to assess the contribution of acceptability and motivational mechanisms in explaining these effects on behavioral measure of PA, physical measures, and health indicators.

One hundred and twenty young women who have undergone BS in the last 3 to 6 months will be included. The volunteers will be randomly assigned to one of three arms: standard care (CONTROL), access to an internet-based physical activity program delivered by an eHealth platform associated with an activity bracelet (ACTI-MOBIL), or access to a physical activity program delivered via videoconferencing (ACTI-VISIO). The primary outcome is the distance traveled during a 6-minute walk test relativized according to Capadaglio's theoretical distance. Secondary outcomes are behavioral measures of physical activity, physical measures, health indicators, technology acceptability, and motivational concepts. Data will be collected baseline (T0), 3 months (T3) and 6 months later (T6). The technology groups will receive a PA program for 12 weeks (between T0 and T3). A mixed model approach will be used to analyze the change in outcomes over time for each group.

This study will provide information on the effects of two technology-based physical activity programs (mobile technology and videoconferencing) after bariatric surgery. Based on the results, recommendations for implementing these programs will be made.

ELIGIBILITY:
Inclusion Criteria:

* Undergone bariatric surgery at a tertial referral center for bariatric surgery (Nice University Hospital, France) 3 to 6 months ago
* Respect with the national recommendations (e.g., BMI ≥ 40kg/m² or ≥ 35kg/m² with at least one co-morbidity among blood hypertension, type 2 diabetes, invalidating arthritis, and sleep apnea syndrome; and no physical disability to practice PA)
* Having a smartphone compatible with the proposed technologies.

Exclusion Criteria:

* Serious adverse events
* Withdrawal of informed consent or violation of the protocol

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Change of functional capacity calculated by the percentage achievement of the theoretical distance calculated by the Capodaglio's (2013) formula | Baseline (T0), 3 months (T3), and 6 months (T6)
  We will aggregate the following primary outcome measures into the Capodaglio (2013) formula: 894.2177 - (2.0700 x age(years)) - (51.4489 x 1) - 5.1663 x BMI (kg/m²) to obtain the theoretical distance, and we will calculate the percentage achievement of this theoretical distance: ((distance traveled(meters) - theoretical distance(meters)) / theoretical distance(meters))x100.
  Higher percentage of achievement reflecting higher functional capacity.
Change of distance traveled during a six-minute walk test (6MWT) | Baseline (T0), 3 months (T3), and 6 months (T6)
  Distance traveled during a six-minute walk test (6MWT) will be expressed in meters
Change of body mass | Baseline (T0), 3 months (T3), and 6 months (T6)
  Kilograms
Height | Baseline (T0)
  Meters
Date of birth | Baseline (T0)
  The date of birth will be requested once (pre-bariatric surgery) and will be used to calculate the age in years at the different periods needed to calculate the theoretical 6MWT distance

SECONDARY OUTCOMES:
Change of subjective physical activity level | Baseline (T0), 3 months (T3), and 6 months (T6)
  Global Physical Activity Questionnaire validated in the French language (Rivière et al., 2018). This scale comprises 16 items to assess the frequency and duration of PA during work, transportation, leisure time, and time spent sitting in a typical week. The items are used to calculate the energy expenditure score in metabolic equivalent tasks (METs), where 150 minutes per week of moderate to vigorous PA corresponds to 600 MET-min/week.
Change of objective physical activity level | Baseline (T0), 3 months (T3), and 6 months (T6)
  Axivity AX3 triaxial accelerometer worn on the wrist during 7-day period. The sensor will be set to begin recording at midnight the day after the appointment over a 7-day period at 100 Hz with a dynamic range of ±8g. The AX3 data will be downloaded, resampled, calibrated and analyzed using open-source AX3 OmGui software (OmGui Version 1.0.0.43, Open Movement, Newcastle University, UK).
Change of stage of change for physical activity | Baseline (T0), 3 months (T3), and 6 months (T6)
  Stage of Change for physical activity will be measured using the French version of the Stages of Change questionnaire (Romain et al., 2012). Regular PA and exercise are defined as "at least 30 minutes per session, at least 5 days per week of moderate to vigorous PA." This questionnaire includes five items with a "yes" or "no" answer, transformed by an algorithm to attribute a score to each participant according to her stage (precontemplation=1, contemplation=2, preparation=3, action=4 or maintenance stage=5).
Change of energetic consumption measured during the 6MWT | Baseline (T0), 3 months (T3), and 6 months (T6)
  The physiological variables will be measured during the 6MWT: oxygen uptake, minute ventilation, carbon dioxide output, respiratory exchange ratio, and heart rate, using the Cosmed K5 system (Cosmed K5, Rome, Italy), which consists of a mask and a portable unit. A decrease in energetic consumption for the same distance travelled during the 6MWT reflecting a better adaptation to exercise.
Change of muscle strength | Baseline (T0), 3 months (T3), and 6 months (T6)
  The maximal isometric knee extensor muscles' strength of the left and right lower limb will be measured with the MicroFET2 (Hoggan Scientific, LLC, Salt Lake City, UT, USA). Women will be seated in a chair with the assessed limb placed at a knee angle of 90° (with full knee extension corresponding to 180°). They will be asked to push as hard as possible for 5 seconds against the dynamometer held by a strap attached to the chair. The highest value in Newton (N) of three measurements will be recorded, and the average of both limbs results will be used for analysis.
Change of quality of life in 5 dimensions | Baseline (T0), 3 months (T3), and 6 months (T6)
  Quality of life will be assessed with the French version of the EuroQoL-5-Dimensions (EQ-5D, Jannssen et al., 2013). The EQ-5D comprises five items measuring quality of life along five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. For each dimension, participants have five response options ranging from "no problems" to "unable." Lower scores indicating better quality of life.
Change of quality of life in visual analog scale | Baseline (T0), 3 months (T3), and 6 months (T6)
  Quality of life will be assessed with the French version of the EuroQoL-visual analog scale (EQ-VAS, Jannssen et al., 2013). The EQ-VAS has a single item for which the women will be asked to rate their current health on a scale from 0: "worst imaginable" to 100: "best imaginable." Higher scores indicating better quality of life
Change of body mass index | Baseline (T0), 3 months (T3), and 6 months (T6)
  Height (meters) and body mass (kilograms) will be measured by medical staff and used to calculate the BMI (kg/m²).
Change of body composition | Baseline (T0), 3 months (T3), and 6 months (T6)
  Body composition will be measured by bioimpedance using the Biody XpertZM (Aminogram, France): muscle mass (kg), fat mass (kg), and bone mineral content (kg). For analyses these measures will be converted to percentages.

OTHER OUTCOMES:
Change of technology acceptability | Baseline (T0), 3 months (T3), and 6 months (T6)
  Measured only in the technologies groups (ACTI-MOBIL, ACTI-VISIO) by the French eHealth acceptability scale (Hayotte et al., 2020). This scale includes 22 items divided into seven subscales: performance expectancy, effort expectancy, social influence, facilitating conditions, hedonic motivation, price value, and habit. Behavioral intention will also be measured using the French translation described in the French eHealth acceptability scale (Hayotte et al., 2020). Participants will rate each item on a 7-point scale ranging from 1: "strongly disagree" to 7: "strongly agree." Higher scores indicating better technology acceptability.
Program compliance | 3 months (T3)
  To measure technology-based program compliance, companies will be asked to report the presence or absence of women and their RPE at each session in a register (directly reported by the PA professional for ACTI-VISIO; completion, content consultation and validation statistics, PA level and number of days the activity bracelet is worn for ACTI-MOBIL).
Change of motivation for physical activity | Baseline (T0), 3 months (T3), and 6 months (T6)
  The motivation for health-oriented PA will be measured with a French motivation scale for health-oriented PA (Boiché et al., 2016). This scale comprises 18 items, equally distributed across the six motivational constructs of self-determination theory: intrinsic motivation, integrated regulation, identified regulation, introjected regulation, external regulation, and amotivation. Participants will respond on a 7-point Likert scale ranging from 1: "strongly disagree" to 7: "strongly agree." Higher scores indicating the most predominant type of motivation on the self-determination continuum.
Change of general causality orientations scale for physical activity | Baseline (T0), 3 months (T3), and 6 months (T6)
  Causality orientations will be measured using an adaptation of the General Causality Orientations Scale (Vallerand et al., 1987) to assess the strength of three motivational orientations (i.e., autonomy, control, impersonal) in the context of PA in a medical environment. The scale comprises seven vignettes and 21 items. Each vignette describes a situation and is followed by three items, one per motivational orientation, to which participants respond on a 7-point scale ranging from 1: "strongly disagree" to 7: "strongly agree." The higher scores indicating the most predominant type of causality orientation.
Change of basic psychological needs | Baseline (T0), 3 months (T3), and 6 months (T6)
  Basic psychological needs will be measured using a French scale validated in the sports context (Gillet et al., 2008) where we replaced "sport" by "physical activity." This scale comprises 15 items distributed across the three needs: autonomy, competence, and relatedness. Participants will respond on a 7-point Likert scale ranging from 1: "strongly disagree" to 7: "strongly agree." The higher scores indicating the most predominant type of basic psychological needs.

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne d'Arripe-Longueville, Pr, Study Director — Université Côte d'Azur, Nice, France
Locations (1):
- Centre Spécialisé Obésité, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hayotte M, Iannelli A, Negre V, Pradier C, Therouanne P, Fuch A, Diagana O, Garbarino JM, Vuillemin A, Colson SS, Chevalier N, d'Arripe-Longueville F. Effects of technology-based physical activity interventions for women after bariatric surgery: study protocol for a three-arm randomised controlled trial. BMJ Open. 2021 Jul 30;11(7):e046184. doi: 10.1136/bmjopen-2020-046184. PMID 34330855